CLINICAL TRIAL: NCT06794320
Title: Antibiotic Stewardship in Suspected Neutropenic Fever (ASTERIC Trial): a Multi-centre, Type 1 Hybrid Effectiveness-implementation, Stepped-wedge, Randomised Controlled Trial
Brief Title: Antibiotic Stewardship in Suspected Neutropenic Fever (ASTERIC Trial)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Prof. Timothy Hudson RAINER, BSc (Hons), MBBCh, MRCP (UK), FHKCEM, FHKAM, MD, FRCEM, FRCP, FIFEM, The University of Hong Kong
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ASTERIC; 21222361 (Other Grant/Funding Number: Health and Medical Research Fund (HMRF))
Record Dates: First submitted 2025-01-14; First posted 2025-01-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2024-10

CONDITIONS: Neutropenic Fever
Keywords: Antibiotic stewardship; Cancer; Carcinoma; Emergency care; Emergency department; Febrile Neutropenia; Health policy; Hematologic Neoplasms; Hospitalization; Length of stay; Meropenem; Neoplasms; Neutrophils; Oncology; Randomized Controlled Trial; RCT; Safety; Tumor
MeSH Terms: conditions — Febrile Neutropenia; Neoplasms; Carcinoma; Emergencies; Hematologic Neoplasms | interventions — NF protocol

STUDY DESIGN:
Masking Description: type 1 hybrid effectiveness-implementation, stepped-wedge, randomised controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Period 1(Before): Standard of Care(SoC) + Neutropenic Fever(NF) Protocol (Other)
  Interventions: Other: NF Protocol
- Period 2(After): SoC + ASTERIC Protocol (Other): The ASTERIC protocol seeks to evaluate and address barriers and facilitators to a fast-track ANC service coupled with prudent, timely antibiotic stewardship and assessment of admission.
  Interventions: Other: ASTERIC protocol

INTERVENTIONS:
Other: NF Protocol — The daily practice of physicians in evaluating and treating patients with sNF.
  Arms: Period 1(Before): Standard of Care(SoC) + Neutropenic Fever(NF) Protocol
Other: ASTERIC protocol — i. Risk-assessment tools
  Arms: Period 2(After): SoC + ASTERIC Protocol
Other: ASTERIC protocol — ii. Fast track absolute neutrophil counts turnaround service
  Arms: Period 2(After): SoC + ASTERIC Protocol
Other: ASTERIC Protocol — iii. A decision tool for patient management and initial antibiotic use
  Arms: Period 2(After): SoC + ASTERIC Protocol
Other: ASTERIC Protocol — iv. A decision tool for patient management and subsequent antibiotic use
  Arms: Period 2(After): SoC + ASTERIC Protocol
Other: ASTERIC Protocol — v. An educational package
  Arms: Period 2(After): SoC + ASTERIC Protocol
Other: ASTERIC Protocol — vi. A decision tool for patient disposal - discharge or emergency department ward observation
  Arms: Period 2(After): SoC + ASTERIC Protocol

SUMMARY:
Executive Summary

Background: Neutropenic Fever (NF), or febrile neutropenia, occurs in patients with early stage and metastatic solid tumours, non-leukaemic haematological cancers and acute leukaemia. It has a crude mortality rate of 3 to 18%. In Hong Kong, and in line with international guidelines, the target time from ED registration to ultra-broad spectrum antibiotic (UBSA) administration (door-to-antibiotic time, DTA time) is one hour disregarding the absolute neutrophil count (ANC). However, over 80% patients presenting to hospital with suspected NF (sNF) do not have NF and do not require UBSAs. Thus there is a need for evidence for a safe role for early treatments in patients with sNF to reduce unnecessary use of antibiotics.

Protocol, Eligibility and Randomisation: This protocol describes the ASTERIC Trial, a pragmatic, multi-centre, type 1, hybrid effectiveness-implementation, stepped-wedge, before and after, cluster randomised controlled trial with variable baseline and follow up periods. Hospitals will be randomised to start dates comparing usual standard of care (SoC) (Period 1, before) with a new antibiotic stewardship protocol (Period 2, after). Hospitals, not patients, are randomised to variable start dates. The evidence for starting early UBSAs in patients with NF is well-established. What is unclear is how to optimise personalised care and the start times of UBSA when the majority of sNF patients do not have NF, there are delays to receiving an ANC report, and a proportion of patients might not need hospital admission.

Study design: a multi-centre, hybrid type 1 effectiveness-implementation trial which is an appropriate study design to evaluate the real-world effectiveness of an antibiotic stewardship protocol; and the barriers to and facilitators of its implementation in the ED setting.

Settings: Eight hospitals in Hong Kong with patient involvement 24/7.

Outcomes: The Trial has two co-primary outcomes 1) mean total dose of UBSAs prescribed in 7 days and censored at 30 days from the time of randomisation; 2) safety (defined as the proportion of patients with a SAE), censored at 30 days from the time of randomisation.

This multifaceted trial addresses three broad domains of implementation according to Proctor's conceptual framework and taxonomy which incorporates the RE-AIM framework, namely: Service Outcomes; Implementation Outcomes and Client outcomes. Simplicity on the frontline: Patient enrolment and other front-line trial procedures will be streamlined. Informed consent is brief and simple and required for follow-up. Follow-up information may be ascertained by contacting participants in person, by phone or electronically, or by review of medical records and databases.

Data to be collected: Information will be collected on the patient, age, sex, major co-morbidity, sNF symptom onset date and severity, as well as any contraindications to study treatments. Follow-up information includes antibiotics - name, dose and duration; SAEs; mortality; sepsis; length of hospital stay; cost-effectiveness; patient satisfaction.

Numbers: 648 patients (324 patients in each group) adult patients with sNF ≥38.3ºC and Modified Early Warning Score ≤6 within 24 hours of ED registration.

Benefit to Healthcare/Expected results: Study results will inform health policy with improvement in hospital services in treating stable sNF evidenced by improved personalised, safe antibiotic stewardship, early antibiotic de-escalation, early discharge, and reduced costs and length of stay. The ASTERIC protocol safely reduces the type, duration and dose of antibiotics.

DETAILED DESCRIPTION:
1 Background and Rationale

1.1 Background

Burden of neutropenic fever Neutropenic fever (NF), or febrile neutropenia, is characterised by a high body temperature and low absolute neutrophil count (ANC) after myelosuppressive cancer treatment. It occurs in patients with early-stage and metastatic solid tumours, non-leukaemic haematological cancers and acute leukaemia. The crude mortality rate varies from 3 to 18%. In the United States (US), each year, 7.83 per 1,000 cancer patients are hospitalised with NF. The mean direct hospitalisation costs of managing NF vary from EUR3,950 [about HKD$ 34,000] to US$19,110 [about HKD$150,000] per patient.

Aetiology

NF can have infectious and non-infectious causes. Although 30 - 50% cases appear clinically to be infections only 20 - 30% have microbiologically documented infections. Bloodstream infections, bacterial translocations from the respiratory tract and perianal region, and from the central venous catheter are major sources.

Fever may be the only manifestation of infection during neutropenia because the typical signs of inflammation are obscured. Neutropenia usually results from myelosuppressive cancer treatments, pre-engraftment phases of haematopoietic stem cell transplantation (HSCT), bone marrow failure and/or defective neutrophil maturation.

Neutropenic Fever

NF is defined by 1) a single oral temperature ≥38.3ºC (101ºF), or a sustained temperature ≥38.0ºC (100.4ºF) over 1 hour; and 2) an ANC <1.0 x 10^9/L ("moderate" neutropenia). Neutropenia is classified as "severe", "profound" or "protracted" if the ANC is 0.5 x 10^9/L, <0.1 x 10^9/L, or lasts for more than one week, respectively. This definition only applies to oncological and haematological patients.

In Hong Kong

Local public emergency departments (EDs) have standard operating procedures and guidelines for managing NF. In line with international guidelines the target time from ED registration to antibiotic administration (door-to-antibiotic time, DTA time) is one hour disregarding ANC. The clinical pathways for suspected NF (sNF) expedites medical consultation, septic workup, and early prescription of ultra-broad spectrum antibiotics (UBSAs) such as Meropenem or Piperacillin/ Tazobactam. After implementing clinical pathways in local EDs, DTA times have shortened.

However, over 80% patients presenting to Hong Kong's Queen Mary Hospital with sNF have an ANC>1x10^9/L, do not have NF, do not require UBSAs and possibly do not require hospital admission. Widespread, inappropriate use of UBSAs may contribute to the emergence of antimicrobial resistance (AMR) and multi-drug resistance strains (MDR). Thus, there is a need for prudent, pragmatic, personalised antibiotic stewardship and appropriate de-escalation.

Antibiotic stewardship for cancer patients

As cancer patients are frequently prescribed antibiotics, they are more vulnerable to MDR, and are in special need of antibiotic stewardship. UBSAs are often started empirically in the ED for patients with sNF, assuming infection by drug-resistant bacteria. However, clinicians infrequently de-escalate once antibiotics have been started. Prolonged exposure to parenteral broad-spectrum antibiotic (BSA) impose risks of nosocomial infection and injection site complications. There is also evidence that meeting the one hour target does not improve outcomes but using appropriate antibiotic regimes does.

Research Gap and Unmet Clinical Need

Evidence-based practices are slow to be implemented into routine care. Implementation science seeks to narrow the research-to practice gap by identifying barriers and facilitators to effective implementation and designing strategies to achieve desired implementation outcomes. Most patients with sNF receive UBSAs. Yet <20% have confirmed NF and 16% have a confirmed microbe. Therefore, it is likely that antibiotics are being used inappropriately. There are knowledge gaps on methods for rapidly delivering ANC results in the acute setting; microbiological patterns (AMR and MDR rates); service, implementation and client outcomes; a lack of understanding on physician and nursing attitudes, perceptions and practice; a lack of good evidence on the real-world effectiveness, safety, and cost-implications of good prescribing practice (antibiotic stewardship and de-escalation); and a need for evidence-based education in patients with sNF. Implementation science supports translational medicine research to practice gaps. It identifies barriers and facilitators to effective implementation and designs evolving strategies to achieve desired service, implementation and client outcomes. This proposal addresses these issues.

1.2 Treatment Strategies

There is good evidence that patients with NF presenting to hospital benefit from early UBSA/BSA treatment and this is reflected in current guidelines. There is also good evidence that patients with NF and a high Multinational Association for Supportive Care in Cancer (MASCC) Risk Index do not need to be admitted to hospital. However, some healthcare settings have adopted a one hour limit on starting BSA/UBSA treatment and admit all patients to hospital. As ANC results are not usually available within one hour, more than 80% sNF may be treated unnecessarily with inappropriate antibiotics. Consequently, there is a need for implementation studies to identify barriers and facilitators of care, and to optimise early management.

There is currently little clinical evidence for the early management of sNF patients presenting to hospital. Early BSA/UBSA is recommended for patients with NF but the evidence for a strict one hour target for the first dose of antibiotics in patients with sNF has little evidence base. Most protocols would not recommend starting antibiotics where they are not necessary.

All patients with sNF will receive SoC during the first period in the participating hospitals. Later, hospitals will switch to the ASTERIC. Initially randomisation will be between hospitals to determine the time that each hospital will convert to the new protocol:

Period 1, Before: Although there is evidence that early treatment of sNF with UBSAs is safe, a high proportion of patients receive antibiotics unnecessarily. Thus, there is uncertainty over implementing personalised care and strategies to optimises antibiotic stewardship.

Period 2, After: The ASTERIC protocol seeks to safely optimise personalised care.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years
* Tympanic temperature ≥38.3ºC within 24 hours before ED registration
* Last chemotherapy or targeted therapy within 6 weeks for any solid tumour, or in any period following therapies against leukaemia, lymphoma, myelodysplastic syndrome, aplastic anaemia, multiple myeloma, or recipient of HSCT.

Exclusion Criteria:

- The decision on how far to apply or deviate from a protocol rests with the clinician. Patients would be excluded from follow up if were unable or unwilling to provide informed consent for data access

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 648 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
7-day mean UBSA dose | Up to 7-days
  Outcome 1 measure: The mean total UBSA dose per patient from ED registration [Continuous]
30-day Severe Adverse Events | Up to 30-days
  Outcome 2 measure: The proportion of patients with an SAE [Binary Y/N]

SECONDARY OUTCOMES:
Mortality | Up to 30-days
  Outcome 3 measure: The proportion of patients with mortality [Binary: Y/N]
Length of Hospital Stay | Up to 30-days
  Outcome 4 measure: Difference in median LOS between period 1 care and period 2 care [Numerical]

OTHER OUTCOMES:
Secondary Service Outcomes: Efficiency | 30-days
  Proportion of eligible patients who receive SoC and ASTERIC Protocol [Binary Y/N]
Safety | 30-days
  Mean of the total number of SAEs per patient who receive SoC and ASTERIC Protocol [Numerical]
Effectiveness in UBSA use | 7-days
  Proportion of patients in each group receiving no UBSAs [Binary Y/N]
Equity | 7-days
  Extent to which the ASTERIC Protocol achieved its goals, reached beneficiaries and addressed specific health needs [Qualitative- Qualitative data from semi- structured interviews]
Staff Satisfaction regarding Patient Centredness | Up to 7-days
  Differentiation of median staff satisfaction score regarding putting the patient first [Score: 0 - 10]
Staff Satisfaction regarding Timeliness | Up to 7-days
  Differentiation of median staff satisfaction score regarding the speed that steps were enacted
Secondary Implementation Outcomes: Acceptability | 7-days
  The perception that the ASTERIC Protocol is agreeable [Numerical Score 0 - 10]
Adoption | 7-days
  The perception that the ASTERIC Protocol employs evidence-based practice [Numerical Score: 0 - 10]
Appropriateness | 7-days
  The perception that the ASTERIC Protocol is a good fit for emergency medicine and ward settings [Qualitative- Qualitative data from semi- structured interviews]
Cost-effectiveness analysis | 7-days
  Cost-effectiveness comparison between SoC and ASTERIC Protocol [Numerical]
  -Incremental cost-effectiveness ratio will be measured in terms of cost per QALY gained, Δcost ASTERIC+SoC / ΔQALY NF+SoC
Feasibility | 7-days
  Perception of the extent to which the ASTERIC Protocol can be carried out in the emergency department and hospital ward [Numerical Score: 0 - 10]
Fidelity | 7-days
  The extent to which the ASTERIC Protocol was carried out in the emergency department and hospital ward [Numerical Score: 0 - 10]
Penetration | 7-days
  The extent to which the ASTERIC Protocol was integrated into the emergency department and hospital ward [Numerical Score: 0 - 10]
Sustainability | 30-days
  The extent to which the ASTERIC Protocol was maintained in the emergency department and hospital ward [Numerical Score: 0 - 10]
Secondary Client Outcomes: Patient Satisfaction | Up to 7-days
  Differentiation of median patient satisfaction score [Score: 0 - 10]
Functional Assessment of Cancer Therapy - General | 30-days
  FACT-G score comparison between the Period 1 care and Period 2 care [Numerical] FACT-G uses a 5-point rating scale (0= Not at all, 1= A little bit, 2= Somewhat, 3= Quite a bit, 4= Very much.)
Functional Assessment of Chronic Illness Therapy - Neutropenia | 30-days
  FACT-N score comparison between the Period 1 care and Period 2 care [Numerical] FACT-N uses a 5-point rating scale (0= Not at all, 1= A little bit, 2= Somewhat, 3= Quite a bit, 4= Very much.)
Functional Assessment of Chronic Illness Therapy - COST | 30-days
  FACIT-COSTS score comparison between the Period 1 care and Period 2 care [Numerical] FACIT-COST uses a 5-point rating scale (0= Not at all, 1= A little bit, 2= Somewhat, 3= Quite a bit, 4= Very much.)
Hospital admission | 30-days
  Proportion of patients admitted to hospital [Binary Y/N]

CONTACTS AND LOCATIONS:
Overall Officials: Professor RAINER Timothy Hudson, MBBCh, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Peyrony O, Gerlier C, Barla I, Ellouze S, Legay L, Azoulay E, Chevret S, Fontaine JP. Antibiotic prescribing and outcomes in cancer patients with febrile neutropenia in the emergency department. PLoS One. 2020 Feb 28;15(2):e0229828. doi: 10.1371/journal.pone.0229828. eCollection 2020. PMID 32109264
- [Background] Freifeld AG, Bow EJ, Sepkowitz KA, Boeckh MJ, Ito JI, Mullen CA, Raad II, Rolston KV, Young JA, Wingard JR; Infectious Diseases Society of America. Clinical practice guideline for the use of antimicrobial agents in neutropenic patients with cancer: 2010 update by the infectious diseases society of america. Clin Infect Dis. 2011 Feb 15;52(4):e56-93. doi: 10.1093/cid/cir073. PMID 21258094
- [Background] Zhu J, Zhou K, Jiang Y, Liu H, Bai H, Jiang J, Gao Y, Cai Q, Tong Y, Song X, Wang C, Wan L. Bacterial Pathogens Differed Between Neutropenic and Non-neutropenic Patients in the Same Hematological Ward: An 8-Year Survey. Clin Infect Dis. 2018 Nov 13;67(suppl_2):S174-S178. doi: 10.1093/cid/ciy643. PMID 30423039
- [Background] Ko HF, Tsui SS, Tse JW, Kwong WY, Chan OY, Wong GC. Improving the emergency department management of post-chemotherapy sepsis in haematological malignancy patients. Hong Kong Med J. 2015 Feb;21(1):10-5. doi: 10.12809/hkmj144280. Epub 2014 Oct 10. PMID 25306894
- [Background] Levy MM, Evans LE, Rhodes A. The Surviving Sepsis Campaign Bundle: 2018 Update. Crit Care Med. 2018 Jun;46(6):997-1000. doi: 10.1097/CCM.0000000000003119. No abstract available. PMID 29767636
- [Background] Taplitz RA, Kennedy EB, Bow EJ, Crews J, Gleason C, Hawley DK, Langston AA, Nastoupil LJ, Rajotte M, Rolston K, Strasfeld L, Flowers CR. Outpatient Management of Fever and Neutropenia in Adults Treated for Malignancy: American Society of Clinical Oncology and Infectious Diseases Society of America Clinical Practice Guideline Update. J Clin Oncol. 2018 May 10;36(14):1443-1453. doi: 10.1200/JCO.2017.77.6211. Epub 2018 Feb 20. PMID 29461916
- [Background] Boxer L, Dale DC. Neutropenia: causes and consequences. Semin Hematol. 2002 Apr;39(2):75-81. doi: 10.1053/shem.2002.31911. PMID 11957188
- [Background] Pizzo PA, Robichaud KJ, Wesley R, Commers JR. Fever in the pediatric and young adult patient with cancer. A prospective study of 1001 episodes. Medicine (Baltimore). 1982 May;61(3):153-65. doi: 10.1097/00005792-198205000-00003. No abstract available. PMID 7078399
- [Background] Pasikhova Y, Ludlow S, Baluch A. Fever in Patients With Cancer. Cancer Control. 2017 Apr;24(2):193-197. doi: 10.1177/107327481702400212. PMID 28441374
- [Background] Kuderer NM, Dale DC, Crawford J, Cosler LE, Lyman GH. Mortality, morbidity, and cost associated with febrile neutropenia in adult cancer patients. Cancer. 2006 May 15;106(10):2258-66. doi: 10.1002/cncr.21847. PMID 16575919
- [Background] Caggiano V, Weiss RV, Rickert TS, Linde-Zwirble WT. Incidence, cost, and mortality of neutropenia hospitalization associated with chemotherapy. Cancer. 2005 May 1;103(9):1916-24. doi: 10.1002/cncr.20983. PMID 15751024
- [Background] Klastersky J, Ameye L, Maertens J, Georgala A, Muanza F, Aoun M, Ferrant A, Rapoport B, Rolston K, Paesmans M. Bacteraemia in febrile neutropenic cancer patients. Int J Antimicrob Agents. 2007 Nov;30 Suppl 1:S51-9. doi: 10.1016/j.ijantimicag.2007.06.012. Epub 2007 Aug 8. PMID 17689933
- [Background] Culakova E, Thota R, Poniewierski MS, Kuderer NM, Wogu AF, Dale DC, Crawford J, Lyman GH. Patterns of chemotherapy-associated toxicity and supportive care in US oncology practice: a nationwide prospective cohort study. Cancer Med. 2014 Apr;3(2):434-44. doi: 10.1002/cam4.200. Epub 2014 Feb 17. PMID 24706592
- [Background] Weycker D, Li X, Edelsberg J, Barron R, Kartashov A, Xu H, Lyman GH. Risk and Consequences of Chemotherapy-Induced Febrile Neutropenia in Patients With Metastatic Solid Tumors. J Oncol Pract. 2015 Jan;11(1):47-54. doi: 10.1200/JOP.2014.001492. Epub 2014 Dec 9. PMID 25491042
- [Derived] Rainer TH, Lam RPK, Tsang TC, Wai AK, Leung SC, Leung RYY, Wong CKH, Gill H, Lam WWT, Wing Lok Chan W, Chi Kin Cheung A, Lau MT, Lee SF, Choi YF, Fong Lun Lee H, Mok KL, Lam HC, Lee SY, Ho Ting Yeung M, Hung IF. Antibiotic stewardship in suspected neutropenic fever (ASTERIC trial): a multicentre, type 1 hybrid effectiveness-implementation, stepped-wedge, randomised controlled trial study protocol. BMJ Open. 2025 Nov 24;15(11):e108010. doi: 10.1136/bmjopen-2025-108010. PMID 41290295